CLINICAL TRIAL: NCT07030790
Title: A Single-center, Randomized, Double-blind, Placebo-Controlled, Dose Escalation, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of a Single Subcutaneous Injection of KLA480 Injection in Healthy Chinese Participants
Brief Title: A Phase I Clinical Study of a Single Dose of KLA480
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KLA480-101
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KLA480 injection 11.3mg (Experimental): 8 subjects receive KLA480 at a dose of 11.3mg and 2 subjects receive the same volume placebo
  Interventions: Drug: KLA480 injection; Drug: Placebo
- KLA480 injection 22.6mg (Experimental): 8 subjects receive KLA480 at a dose of 22.6mg and 2 subjects receive the same volume placebo
  Interventions: Drug: KLA480 injection; Drug: Placebo

INTERVENTIONS:
Drug: KLA480 injection — Subcutaneous injection，Single dose
Drug: Placebo — Subcutaneous injection，Single dose

SUMMARY:
Primary purpose:

To evaluate the safety and tolerability of KLA480 injection after a single subcutaneous injection in healthy participants.

Secondary purpose:

To evaluate the pharmacokinetic (PK) characteristics of KLA480 injection after a single subcutaneous injection in healthy participants.

DETAILED DESCRIPTION:
This study was a single-center, randomized, double-blind, placebo-controlled, dose Escalation, phase I clinical study to evaluate the safety, tolerability and pharmacokinetic characteristics of KLA480 injection after a single subcutaneous injection in healthy Chinese participants.

The plan is to enroll 20 healthy participants in two dose groups: Group I (11.3 mg) and Group II (22.6 mg). Each dose group will includ 10 participants (at least 3 single-sex participants). Among them, 8 participants received the experimental drug KLA480 injection, and 2 participants received the placebo KLA480 injection simulator. Participants in different dose groups were successively enrolled. Based on the evaluation of acceptable tolerance and safety of participants in the former dose group, the researchers will discuss with the sponsor whether to carry out the next dose group. The "sentinel" method was used in each dose group, that is, 3 participants were enrolled in each dose group first, of which 2 participants received KLA480 injection, and 1 participant received placebo KLA480 injection simulator. Tolerance assessment will be performed 48 h after administration of the first 3 participants, and if the tolerance evaluation is acceptable, the remaining 7 participants in the current dose group will be enrolled (6 receiving the experimental drug and 1 receiving placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Participants could understand and abide by the study process, voluntarily participate in the study, and sign the informed consent form in person;
2. Healthy adult participants of both sexes aged 18 to 45 years (including boundary values);
3. A body weight of at least 50.0 kg for men and 45.0 kg for women. BMI in the range of 18.0-28.0 kg/m2 (including the boundary value);
4. The results of vital signs, physical examination, laboratory examination, chest X-ray (anteroposterior), and electrocardiogram were normal or abnormal with no clinical significance judged by the investigators;
5. Any female or male participant of potential fertility must agree not to donate sperm or eggs from the date of sign informed consent form until 3 months after the last dose, must use an effective contraceptive method, and before the last visit，participants must use nonpharmacologic contraceptive methods to prevent pregnancy or to impregnate a partner.

Exclusion Criteria:

1. Participants with a history of severe allergy or allergy to any component or vehicle components of rotigotin or other non-ergotamine dopamine agonists (pramipexole, ropinirole, piribedil, and apomorphine) ;
2. Participants with a history of gastrointestinal, renal, hepatic, neurological, hematologic, endocrine, tumor, pulmonary, immune, psychiatric, or cardio-cerebrovascular diseases with clinical significance judged by the investigators;
3. History of unexplained orthostatic hypotension, syncope or low systolic blood pressure;
4. Participants with a history of acute infection or other acute diseases within 2 weeks before signing the informed consent form;
5. Those who had unprotected sexual behavior within 2 weeks before signing the informed consent form;
6. Participants who cannot tolerate venous puncture or have a history of fainting blood or fainting needles;
7. Donating blood or massive blood loss (≥400 mL), or receiving blood transfusion/use of blood products within 3 months before signing the informed consent form;
8. Participants who had undergone surgery that would affect the absorption, distribution, metabolism, or excretion of drug as judged by the investigators within 6 months before signing the informed consent form, or had undergone surgery within 4 weeks before the first dose of the trial drug, or planned to undergo surgery between signing the informed consent form and the last visit;
9. Participated in any drug/device clinical trial and used the experimental drug/device within 3 months before signing the informed consent form;
10. Those who had been vaccinated within 1 month before signing the informed consent form, or planned to be vaccinated between signing the informed consent form and the last visit;
11. Strong or moderate inhibitors and/or inducers of liver metabolic enzymes (CYP1A2, CYP2C19, CYP3A4) of rotigotin was using within 4 weeks before the first dose of the trial drug. Examples: Fluvoxamine, Fluconazole, Fluoxetine, ticlopidine, Ceritinib, atanavir, Adrasib, telithromycin, Clarithromycin, itraconazole, ketoconazole, posaconazole, voriconazole, indinavir, Nefinavir, ritonavir, Saquinavir, telanavir, Lopinavir, Nefaketozole, Cobirestat, Apalutamide, enzalutamide, Lumacato, Mitol Tam, ivoclib, phenytoin, carbamazepine, rifampicin, St John's wort;
12. Who used any prescription drug, over-the-counter drug, vitamin product or Chinese herbal medicine within 2 weeks before the first dose of the trial drug;
13. During the screening period, systolic blood pressure decreased ≥20 mmHg or diastolic blood pressure decreased ≥10 mmHg within 3 minutes from supine to upright position, or supine systolic blood pressure < 100 mmHg;
14. Participants with QTcF > 450 ms during the screening period;
15. Hepatitis B virus surface antigen, hepatitis C virus antibody, TPPA antibody, human immunodeficiency virus antibody test results are positive;
16. Female participants with positive pregnancy results or in the lactation period;
17. Had a history of drug abuse or drug use within 6 months before signing the informed consent form, or had a positive result of urine drug screening;
18. Had a history of heavy drinking within 6 months before signing the informed consent form (heavy drinking was defined as drinking 14 units of alcohol per week: 1 unit = beer 285 mL, or spirits 25 mL, or wine 100 mL), or could not give up drinking from signing the informed consent form to the last visit, or had a positive result of alcohol breath test;
19. Participants who had smoked more than 3 cigarettes per day within 3 months before signing the informed consent form, smoked or used tobacco products within 2 weeks before the first dose of the trial drug, or could not give up smoking between signing the informed consent form and the last visit, or had a positive result of tobacco screening test;
20. Participants who consumed grapefruit or a drink containing grapefruit juice within 2 weeks before the first dose of the trial drug;
21. Those who consumed chocolate, any food or drink containing caffeine (such as coffee, tea, milk tea, cola, red bull, etc.) or rich in xanthine (such as shiitake mushroom, silver carp, mulberry, seafood (silver beetle, white hairtail, oyster, white pomade, eel, etc.), animal organs (duck liver, chicken liver, pig large intestine, pig liver, beef liver, etc.) within 72 hours before the first dose of the trial drug;
22. Those who have special dietary requirements and cannot follow the uniform diet during hospitalization;
23. Participants with other factors considered by the investigator to be ineligible for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Collected from signing of informed consent until 43 days after a single dose.
  Safety and tolerability was assessed by the number of participants with adverse events (AE).

SECONDARY OUTCOMES:
Maximum peak plasma concentration (Cmax) [Pharmacokinetics] | 43 days after a single dose.
  Samples will also be collected until 43 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
Time of Cmax (tmax) [Pharmacokinetics] | 43 days after a single dose.
  Samples will also be collected until 43 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
Area under the concentration-time curve (AUC) from time zero to time "t" [Pharmacokinetics] | 43 days after a single dose.
  Samples will also be collected until 43 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
AUC from time zero to infinity (AUC∞) [Pharmacokinetics] | 43 days after a single dose.
  Samples will also be collected until 43 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
Terminal-phase elimination half-life (t1/2,z) [Pharmacokinetics] | 90 days after a single dose.
  Samples will also be collected until 43 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No